CLINICAL TRIAL: NCT04447638
Title: Percutaneous Tracheostomy With Aerosol Box in COVID-19 Positive Patients in Intensive Care Unit: a Clinical Trial
Brief Title: Percutaneous Tracheostomy With COVID-19
Status: Completed | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Mesut ERBAS, Associate Professor, Çanakkale Onsekiz Mart University
Other Study IDs: TT17
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Tracheostomy
Keywords: Reanimation
MeSH Terms: interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tracheostomy with aerosol box in COVID-19 positive patients — Patients who underwent percutaneous tracheostomy with aerosol box in COVID-19 positive patients. The patients age, gender, hospitalization diagnosis, number of intubated days, anesthetic agents used during the procedure, neck ultrasonography data before and during the procedure, and complications were recorded.

SUMMARY:
Coronavirus disease 2019 (COVID-19) has brought about a requirement of intensive care and mechanical ventilation for a significant portion of patients. Percutaneous tracheostomy is performed in order to reduce the complications that may develop due to prolonged endotracheal intubation.

DETAILED DESCRIPTION:
Different methods are needed for situations in which the potential for producing aerosols is high, such as intubation and tracheostomy. One of these methods is the aerosol box.To share our experiences of percutaneous tracheostomy performed with aerosol box in COVID-19 patients. Patients who underwent percutaneous tracheostomy between March 2020 and June 2020 in the pandemic intensive care unit were evaluated retrospectively.The study is designed as a clinical trial study. This study was performed in faculty of medicine hospital's intensive care unit which is located in Canakkale province Turkey.

ELIGIBILITY:
Inclusion Criteria:

* who underwent percutaneous tracheostomy with COVID-19(+)

Exclusion Criteria:

* Patients who do not give informed consent or do not want to participate in the study
* Coagulopathy, thrombocytopenia

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Percutaneous tracheostomy performed with aerosol box in COVID-19 patients
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Complications observed in the cases in which we applied percutaneous tracheostomy with aerosol box | During the procedure
  Complications

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided